CLINICAL TRIAL: NCT02732327
Title: A Single-Center, Randomized, Open-label, Prospective, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftazidime-Avibactam (CAZ-AVI) Plus Vancomycin or Linezolid Versus Standard of Care Plus Vancomycin or Linezolid as Empiric Therapy in Febrile Neutropenic Adults With Cancer
Brief Title: Comparative Study of Ceftazidime-Avibactam Versus Standard of Care as Therapy in Febrile Neutropenic Adults With Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer aligned with the revised clinical development plan and commercial strategy
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAZ-MD-13
Record Dates: First submitted 2016-03-18; First posted 2016-04-08 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Neoplasms; Febrile Neutropenia
MeSH Terms: conditions — Neoplasms; Febrile Neutropenia | interventions — Vancomycin; Linezolid; Cefepime; Meropenem; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAZ-AVI + Vancomycin or Linezolid (Experimental): Ceftazidime-Avibactam (CAZ-AVI) 2.5 mg intravenous (IV) infusion every 8 hours for 5 to 14 days, duration determined by the investigator, plus vancomycin 15 mg/kg IV or linezolid 600 mg IV every 12 hours. A switch to open-label oral or IV therapy (IV therapy for outpatient or home administration per local standard of care [SOC]) may be allowed after at least 72 hours (ie, minimum of 9 doses for CAZ-AVI) of inpatient IV study drug.
  Interventions: Drug: CAZ-AVI; Drug: Vancomycin; Drug: Linezolid
- Standard of Care+Vancomycin or Linezolid (Active Comparator): Standard of Care (cefepime 2 g IV infusion every 8 hours or meropenem 1 g IV infusion every 8 hours or piperacillin/tazobactam 4.5 g IV infusion every 6 hours for 5 to 14 days, duration determined by the investigator) plus vancomycin 15 mg/kg IV or linezolid 600 mg IV every 12 hours. A switch to open-label oral or IV therapy (IV therapy for outpatient or home administration per local SOC) may be allowed after at least 72 hours (ie, minimum of 9 doses for SOC therapies, except piperacillin/tazobactam, which is a minimum of 12 doses) of inpatient IV study drug.
  Interventions: Drug: Vancomycin; Drug: Linezolid; Drug: Cefepime; Drug: Meropenem; Drug: Piperacillin/tazobactam

INTERVENTIONS:
Drug: CAZ-AVI — Ceftazidime-Avibactam (2 g ceftazidime and 0.5 g avibactam)
  Arms: CAZ-AVI + Vancomycin or Linezolid
Drug: Vancomycin — 15 mg/kg
  Other Names: Vancocin
Drug: Linezolid — 600 mg
  Other Names: Zyvox
Drug: Cefepime — 2 g
  Other Names: Maxipime
  Arms: Standard of Care+Vancomycin or Linezolid
Drug: Meropenem — 1 g
  Other Names: Merrem
  Arms: Standard of Care+Vancomycin or Linezolid
Drug: Piperacillin/tazobactam — 4.5 g
  Other Names: Zosyn
  Arms: Standard of Care+Vancomycin or Linezolid

SUMMARY:
This study will evaluate the effect, safety, and tolerability of ceftazidime-avibactam (CAZ-AVI) plus vancomycin or linezolid compared to standard of care plus vancomycin or linezolid as empiric therapy in febrile neutropenic adults with cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with neutropenic fever who have existing malignancy or have undergone hematopoietic stem cell transplantation
* Requires hospitalization for intravenous (IV) empiric antibiotic therapy

Exclusion Criteria:

* Fungal or viral infection requiring additional therapy
* Known acute viral hepatitis
* Known to be human immunodeficiency virus (HIV) positive
* Expected requirement for hemodialysis while on study therapy
* Received >24 hours of systemic antibacterial therapy within 72 hours of initiation of inpatient IV study drug
* Past or current history of epilepsy or seizure disorder
* Evidence of immediately life-threatening disease, progressively fatal disease, or life expectancy of 3 months or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, M.D., Study Director — Allergan
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned sample size was 100 patients; however, the sponsor discontinued the study due to the fact that the study no longer aligned with the revised clinical development plan and commercial strategy for CAZ-AVI. A total of 2 patients were enrolled and completed the study.
Period: Overall Study
Arm/Group | CAZ-AVI + Vancomycin or Linezolid | Standard of Care+Vancomycin or Linezolid
Started | 0 | 2
Completed | 0 | 1
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAZ-AVI + Vancomycin or Linezolid | Standard of Care+Vancomycin or Linezolid | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years |  | 2 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Favorable Clinical Response at End of Inpatient Intravenous Therapy (EOIV)
Description: Favorable clinical response is defined as resolution of all acute signs and symptoms of the primary infection or improvement to such an extent that no additional antibacterial therapy is required as assessed by the investigator. Due to study termination and limited enrollment, outcome measures were not analyzed.
Time Frame: Up to Day 14
Arm/Group | CAZ-AVI + Vancomycin or Linezolid | Standard of Care+Vancomycin or Linezolid
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Due to termination of the study, adverse events were not coded.
Arm/Group | CAZ-AVI + Vancomycin or Linezolid | Standard of Care+Vancomycin or Linezolid
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAZ-AVI + Vancomycin or Linezolid (N=0) | Standard of Care+Vancomycin or Linezolid (N=2)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.